CLINICAL TRIAL: NCT06658262
Title: Effects Of Tai Chi Exercises With Cycling Exercises On Balance, Gait And Quality Of Life In Sub-Acute Stroke Patients
Brief Title: Effects of Tai Chi Exercises With Cycling in Subacute Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0209
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Stroke
Keywords: CVA,; Tai Chi; Stroke; Rehabilitation; Gait Parameters; Cycling
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Tai Chi Exercises + Cycling exercises. Treatment session of 60 min will be given 3 times a week for 6 weeks.
  Interventions: Other: Tai Chi Exercises With Cycling Exercises
- Control Group (Other): Tai Chi Exercises Alone. Treatment session of 60 min will be given 3 times a week for 6 weeks.
  Interventions: Other: Tai Chi Exercises Alone

INTERVENTIONS:
Other: Tai Chi Exercises With Cycling Exercises — Tai Chai exercises include Ward Off: This movement involves extending and redirecting energy, promoting stability and balance through controlled shifts in weight and posture. Grasp Sparrow's Tail: It comprises a series of movements that emphasize weight shifting, coordination, and maintaining a stable stance, all of which contribute to improved balance and gait. 3.Single Whip: This movement focuses on shifting weight smoothly from one foot to the other while maintaining proper alignment, helping to enhance proprioception and stability. 4.Brush Knee and Twist Step: By incorporating controlled twists and steps, this movement helps to improve coordination, strengthen leg muscles, and refine gait dynamics. Participants will be assisted to safely mount the ergometer bicycle. The height of the seat will be adjusted to ensure postural balance, upright seating and firm contact of the feet with the pedals. Treatment for the cycling will last for 30 minutes per session.
  Arms: Experimental Group
Other: Tai Chi Exercises Alone — Tai Chai exercises include Ward Off: This movement involves extending and redirecting energy, promoting stability and balance through controlled shifts in weight and posture. Grasp Sparrow's Tail: It comprises a series of movements that emphasize weight shifting, coordination, and maintaining a stable stance, all of which contribute to improved balance and gait. 3.Single Whip: This movement focuses on shifting weight smoothly from one foot to the other while maintaining proper alignment, helping to enhance proprioception and stability. 4.Brush Knee and Twist Step: By incorporating controlled twists and steps, this movement helps to improve coordination, strengthen leg muscles, and refine gait dynamics. 5.Part the Wild Horse's Mane
  Arms: Control Group

SUMMARY:
Stroke, a debilitating cerebrovascular event, frequently leads to severe motor and sensory impairments resulting in a diminished quality of life. Tai Chi, an ancient Chinese martial art known for its slow, flowing movements, emphasis on breath control, and mindfulness, presents an intriguing avenue for stroke rehabilitation. While cycling exercises facilitates muscle control of the lower limbs, which may allow putting more weight on the affected leg while standing, also beneficial for stroke survivors.

DETAILED DESCRIPTION:
This is two-arm parallel design randomized controlled trial. Participants will be selected by non-probability consecutive sampling technique, fifty stroke patients meeting the inclusion criteria will be randomly allocated into two groups (experimental and control) by online randomizer tool. The experimental group will receive tai chi exercises with cycling exercises and the control group will receive tai chi exercises alone. Treatment session of 60 min will be given 3 times a week for 6 weeks. The following primary and secondary assessment tools will be used, Functional Reach Test and Berg Balance scale for balance, Dynamic Gait Index and Wisconsin Gait Scale for gait assessment and Stroke Specific Quality of life (SS-QOL). The data will be analyzed using SPPS software version. 26.

ELIGIBILITY:
Inclusion Criteria:

* Participants with the age ranged between 50-65 years.
* Participants with either gender.
* Patients who are in the sub-acute phase (from 2 weeks to less than 3 months after onset).
* No visual field defect.
* No abnormality of the vestibular organs.
* No orthopedic disease.
* The ability to understand and perform the exercise as instructed by the researcher
* Muscle power of at least grade three.
* Could walk at least 10 meters with or without assistive devices.

Exclusion Criteria:

* Chronic stroke patient.
* Participants with aphasia and cognitive impairment.
* Cardiac arrhythmias
* Any condition for which exercise is contraindicated
* Fracture of the lower limb.
* Participants who are currently participating in another clinical trial or research study.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-24 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-02-03 (Estimated)

PRIMARY OUTCOMES:
Dynamic Gait Index | 6 weeks
  The DGI is developed to assess the likelihood of falling in older adults. It is designed to test eight facets of gait. Equipment needed: Box (Shoebox), Cones (2), Stairs, 20' walkway, 15" wide. Completion time is 15 minutes. A four-point ordinal scale, ranging from 0-3 is used for scoring. "0" indicates the lowest level of function and "3" the highest level of function. Total Score = 24. The ICC2 for intra-rater and inter-rater reliability of total DGI scores is 0.86 and 0.91 respectively.
Berg Balance Scale | 6 Weeks
  Balance will be measured using the Berg Balance Scale (BBS).The BBS is a 14-item scale that quantitatively assesses balance through direct observations of the performance ability, with each item scored from 0 ('inability to complete the task') to 4 ('independent completion'). The total possible score is 56 points, with higher scores indicating that the person has better balance. The berg balance scale reliability is 0.98, validity: r=0.91
Stroke Specific Quality Of Life (SS-QOL): | 6 weeks
  The perceived QOL will be measured using the Korean version of the Stroke-Specific Quality of Life questionnaire (SS-QOL), which evaluates the level of energy, family roles, language, mobility, mood, social roles, personality, thinking, and self-care using a 5-point Likert scale. The validity of psychometrics measures of the original version of the scale was reported, with a reliability coefficient of 0.73-0.89. Cronbach's values for the subscales of the SS-QOL were 0.92-0.93 among stroke survivors.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Asrar Yousaf, Mphil, Principal Investigator — Riphah International University
Locations (1):
- Ittefaq Hospital Lahore., Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jing C, Li K, Li Z, Sun Y, Wu J, Li Y, Li Y, Zhou L, Zhang Z, Zhao M, Zhang Y. Tai Chi postural training for dyskinesia rehabilitation: a study protocol for a randomised controlled trial in convalescent ischaemic stroke patients. BMJ Open. 2021 May 18;11(5):e046003. doi: 10.1136/bmjopen-2020-046003. PMID 34006551
- [Background] Hsu CY, Moyle W, Cooke M, Jones C. Seated Tai Chi versus usual activities in older people using wheelchairs: A randomized controlled trial. Complement Ther Med. 2016 Feb;24:1-6. doi: 10.1016/j.ctim.2015.11.006. Epub 2015 Dec 2. PMID 26860794
- [Background] Thant AA, Wanpen S, Nualnetr N, Puntumetakul R, Chatchawan U, Hla KM, Khin MT. Effects of task-oriented training on upper extremity functional performance in patients with sub-acute stroke: a randomized controlled trial. J Phys Ther Sci. 2019 Jan;31(1):82-87. doi: 10.1589/jpts.31.82. Epub 2019 Jan 29. PMID 30774211
- [Background] Batool S, Zafar H, Gilani SA, Ahmad A, Hanif A. Intrarater and interrater reliability of the dynamic gait index in post stroke patients with eye movement disorders. J Bodyw Mov Ther. 2023 Jul;35:38-42. doi: 10.1016/j.jbmt.2023.04.015. Epub 2023 Apr 14. PMID 37330797
- [Background] Perez-de la Cruz S. Comparison between Three Therapeutic Options for the Treatment of Balance and Gait in Stroke: A Randomized Controlled Trial. Int J Environ Res Public Health. 2021 Jan 7;18(2):426. doi: 10.3390/ijerph18020426. PMID 33430476